CLINICAL TRIAL: NCT00484159
Title: Prospective Randomized Study Comparing 0, 1, and 2 Diagnostic Lumbar Medial Branch (Facet Joint) Blocks Before Radiofrequency Denervation in Patients With Chronic Low Back Pain: A Cost: Benefit Analysis.
Brief Title: Efficacy and Cost: Benefit Ratio of 0, 1, and 2 Medial Branch Blocks for Lumbar Facet Joint Radiofrequency Denervation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Office of Research Administration, Amanda Gibson
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00007158
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2009-01

CONDITIONS: Low Back Pain
Keywords: Low back pain of suspected lumbar zygapophysial etiology
MeSH Terms: conditions — Low Back Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Radiofrequency lumbar facet joint denervation only if positive response to 2 diagnostic facet blocks.
  Interventions: Procedure: Radiofrequency denervation of medial branches; Drug: 0.5% bupivacaine; Drug: 2% lidocaine; Procedure: Radiofrequency denervation
- 2 (Experimental): Radiofrequency lumbar facet joint denervation if positive response to single facet joint block.
  Interventions: Procedure: Radiofrequency denervation of medial branches; Drug: 0.5% bupivacaine; Procedure: Radiofrequency denervation
- 3 (Experimental): Radiofrequency lumbar facet denervation without a diagnostic facet block.
  Interventions: Procedure: Radiofrequency denervation of medial branches; Procedure: Radiofrequency denervation

INTERVENTIONS:
Procedure: Radiofrequency denervation of medial branches — Radiofrequency of medial branches that innervate the lumbar facet joints
Drug: 0.5% bupivacaine — Diagnostic medial branch block with 0.5% bupivacaine. Blocking the nerves that innervate the facet joints with a long-acting local anesthetic.
  Arms: 1; 2
Drug: 2% lidocaine — Diagnostic medial branch block with 2% lidocaine. Blocking the nerves that innervate the facet joints with a short-acting local anesthetic.
  Arms: 1
Procedure: Radiofrequency denervation — Radiofrequency lumbar facet denervation without a diagnostic block
  Arms: 3
Procedure: Radiofrequency denervation — Radiofrequency lumbar facet denervation only if positive response to 2 diagnostic blocks.
  Arms: 1
Procedure: Radiofrequency denervation — Lumbar facet radiofrequency denervation if positive response to a single diagnostic facet block
  Arms: 2
Procedure: Radiofrequency denervation — Radiofrequency lumbar facet denervation without a diagnostic facet block.
  Arms: 3

SUMMARY:
Lumbar zygapophysial (facet) joint pain is a common cause of low back pain. Radiofrequency (RF) denervation is an effective and low risk treatment of chronic low back pain of suspected facet joint etiology. Blocks of the medial branches innervating the joints are commonly used to localize the pain and make the diagnosis of facet joint pain.

There is currently no standard number of diagnostic blocks: zero, one, and two blocks have all been utilized. Considering the high false positive and false negative rates of these blocks, the cost: benefit ratio has been questioned. No study to date has examined the practice of diagnostic medial branch blocks before RF denervation.

The purpose of this study is to determine the optimal number of blocks before radiofrequency denervation. Three groups of patients will be studied. In group I, patients will undergo RF denervation based on history and physical exam alone. In group II, patients will undergo RF denervation based on a positive response to a single diagnostic block with local anesthetic. In group III, patients will undergo RF treatment only after a positive screening block and a positive confirmatory block.

DETAILED DESCRIPTION:
Lumbar zygapophysial (facet) joints are recognized as one of the most common causes of chronic low back pain with an estimated prevalence among patients with LBP ranging from 15% to 40%. Radiofrequency (RF) denervation of facet joints has been utilized as an effective treatment of chronic pain attributed to these joints. Blocks of the medial branches innervating the joints are commonly used to localize the pain and make a diagnosis of lumbar zygapophysial (l-z) joint pain. However, considering the high false-positive rates of these blocks (25-40%), the false-negative rates (8-10%), and the number of blocks necessary to make the diagnosis before treatment, the cost-effectiveness of performing these blocks and the benefit of exposing these patients to additional risks is under question. The risks of RF denervation are so low (equivalent to performing the diagnostic block), some have questioned whether or not any diagnostic facet blocks should be performed before RF lesioning.

The purpose of the study is to determine the optimal number of diagnostic blocks that should be performed before radiofrequency denervation in patients with chronic lower back pain with suspected facet joint etiology.

In this prospective randomized study, we will recruit 150 patients with suspected chronic (l-z) joint pain without neurological symptoms to undergo one of three treatment modalities. In group I, 50 patients will undergo RF denervation based on history and physical exam alone (what we advocate in a recent review article). In group II, 50 patients will receive a single diagnostic block with 0.5% bupivacaine. Those that obtain greater than 50% pain reduction will undergo RF denervation. In group III, 50 patients will receive a block with either 2% lidocaine or 0.5% bupivacaine. Those patients that obtain greater than 50% pain relief with the first block receive a second block with the other local anesthetic. Patients that obtain greater than 50% pain relief with the second block then undergo RF. Patients in any group that obtain less than 50% pain relief with any block exit the study.

ELIGIBILITY:
Inclusion Criteria:

* Axial low back pain unresponsive to conservative treatment measures such as physical therapy, manual therapy and pharmacotherapy
* Duration of pain greater than 6 months

Exclusion Criteria:

* Age younger than 18 years
* Objective evidence (MRI or physical exam findings) of lumbosacral radiculopathy
* Prior radiofrequency treatment
* Significant spinal stenosis or spondylolisthesis
* Previous back surgery
* Uncorrected coagulopathy
* Unstable medical or psychiatric condition
* Pregnancy
* Allergies to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins School of Medicine, Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 patients with axial low back pain and suspected lumbar facet arthropathy were recruited from pain clinics at Johns Hopkins and Walter Reed between January 2007 and April 2009 for lumbar facet interventions.
Pre-assignment Details: Subjects had to be candidate for facet blocks or radiofrequency denervation. They had to have no neurological symptoms, failed conservative treatment and not had spinal fusion.
Groups:
- Double-block Group: Radiofrequency lumbar facet joint denervation only if positive response to 2 diagnostic facet blocks.
- Single-block Group: Radiofrequency lumbar facet joint denervation if positive response to single facet joint block.
- Radiofrequency Group: Radiofrequency lumbar facet denervation without a diagnostic facet block.
Period: Overall Study
Arm/Group | Double-block Group | Single-block Group | Radiofrequency Group
Started | 50 | 50 | 51
Completed | 49 | 49 | 51
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-block Group | Single-block Group | Radiofrequency Group | Total
Number analyzed (Participants) | 50 | 50 | 51 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 45 | 133
  >=65 years | 6 | 6 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 20 | 67
  Male | 27 | 26 | 31 | 84

OUTCOME MEASURES:

1. Primary Outcome: Cost Per Successful Procedure
Description: Total cost per effective treatment at 3-months. Successful procedure defined as greater or equal to 50% pain relief and satisfaction lasting at least 3 months.
Time Frame: 3-months
Measure: Number; unit: U.S. dollars
Arm/Group | Double-block Group | Single-block Group | Radiofrequency Group
Number analyzed (Participants) | 50 | 50 | 51
U.S. dollars | 15,241 | 17,142 | 6286

2. Secondary Outcome: Successful Treatment
Description: Greater or equal to 50% pain relief plus procedural satisfaction lasting at least 3 months. What is being measured is the number of participants with a positive outcome.
Time Frame: 3-months postprocedure
Measure: Number; unit: participants
Arm/Group | Double-block Group | Single-block Group | Radiofrequency Group
Number analyzed (Participants) | 50 | 50 | 51
participants | 9 | 7 | 17

ADVERSE EVENTS:
Arm/Group | Double-block Group | Single-block Group | Radiofrequency Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/51

LIMITATIONS AND CAVEATS:
This study only followed patients for 3 months, so we don't know if proceeding straight to radiofrequency is associated with the same duration of pain relief as when diagnostic facet blocks are performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No